CLINICAL TRIAL: NCT03516357
Title: Effects on Ocular Parameters of Myopic Eyes After Orthokeratology in Myopic
Brief Title: Effects on Ocular Parameters of Myopic Eyes After Orthokeratology in Myopic Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Other Study IDs: YFZX2017002
Record Dates: First submitted 2018-04-12; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2017-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- low myopia: -3.00D < spherical equivalent refractive error < -0.50D
- moderate myopia: -6.00D < spherical equivalent refractive error ≤ -3.0D
- high myopia: spherical equivalent refractive error ≤ -6.0D

SUMMARY:
Effects on Ocular Parameters of Myopic Eyes After Orthokeratology in Myopic Children

DETAILED DESCRIPTION:
1.The primary objective of the current study is to investigate changes in uncorrected visual acuity, diopter, accommodation, peripheral refraction, IOP, tear film quality, corneal thickness, corneal topography, corneal biomechanical parameters, objective optical quality, corneal and conjunctiva sensitivity and choroidal thickness for children with different diopters after wearing orthokeratology lenses; 2. Through measure long-term changes of these parameters, including corneal topography, axial length, peripheral refraction, objective optical quality and choroidal thickness, to explore occurrence and development regularity of myopia.

ELIGIBILITY:
Inclusion Criteria:

* 1. subjects were 6-16 years of age; 2.had no other ocular diseases aside from refractive error and no keratoconus (confirmed by pre-treatment corneal topography); 3. had an intraocular pressure (IOP) of <21 mmHg; 4. had an with-the- rule astigmatism (axes 180 ± 30) ≤ 1.50 D; 5.had a best corrected visual acuity（BCVA） ≤0.00 log MAR units in both eyes (Snellen equivalent to 20/20);

Exclusion Criteria:

* 1. had binocular vision problems; 2.use medications that might affect refractive development; 3.had history of ortho-k or contact lens wear; 4. Ocular surface diseases and other eye diseases which can cause abnormalities of ocular surface; 5. Patients with histories of ocular injury or surgery; 6. Corneal staining and decentration of lens after wearing Ortho-k.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: myopia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2022-01-11 (Estimated); Study Completion 2022-01-11 (Estimated)

PRIMARY OUTCOMES:
axial length measured by IOL-master | 2 years
  measured by IOL-master

SECONDARY OUTCOMES:
accommodation measured by open field auto ref/keratometer measurements(WAM-5500,Grand Seiko) | 2 years
  measured by open field auto ref/keratometer measurements(WAM-5500,Grand Seiko)
peripheral refraction measured by open field auto ref/keratometer measurements(WAM-5500,Grand Seiko) | 2 years
  measured by open field auto ref/keratometer measurements(WAM-5500,Grand Seiko)
IOP measured by Corvis-ST | 2 years
  measured by Corvis-ST
corneal thickness measured by Corvis-ST | 2 years
  measured by Corvis-ST
corneal biomechanical parameters measured by Corvis-ST | 2 years
  measured by Corvis-ST
tear film quality measured by Keratography | 2 years
  measured by Keratography
corneal morphological characteristics measured by Optikon 2000 corneal topographer | 2 years
  measured by Optikon 2000 corneal topographer
objective optical quality measured by OQAS visual quality analyzing system | 2 years
  measured by OQAS visual quality analyzing system
corneal and conjunctiva sensitivity measured by Cochet-Bonnet | 2 years
  measured by Cochet-Bonnet
choroidal thickness measured by ocular coherence tomography | 2 years
  measured by ocular coherence tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Jingan, China

IPD SHARING:
Plan to Share IPD: Undecided